CLINICAL TRIAL: NCT01485809
Title: A Phase II Trial of Gefitinib in Squamous NSCLC Patients Who Failed First-Line Chemotherapy
Brief Title: Efficacy and Safety Study of Gefitinib in Squamous NSCLC Patients Who Failed First-Line Chemotherapy
Acronym: SIIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul Veterans Hospital (Other)
Responsible Party: Principal Investigator, Bong-Seog Kim, Principal investigator, Seoul Veterans Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SVH-1
Record Dates: First submitted 2011-11-24; First posted 2011-12-06 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Squamous Cell Carcinoma of Bronchus
MeSH Terms: interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gefitinib (Experimental)
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — Gefitinib 250mg/day, oral daily q every 4 weeks
  Other Names: Iressa

SUMMARY:
Gefitinib was the first epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) approved for the treatment of advanced non-small cell lung cancer (NSCLC). Results from two randomised phase II trials (IDEAL 1 and 2) suggested that gefitinib was efficacious and less toxic, compared with previous results, than was chemotherapy in patients with previously-treated non-small-cell lung cancer. Two phase III trials of gefitinib in advanced non-small-cell lung cancer followed on from the IDEAL phase II studies: Iressa Survival Evaluation in Lung cancer (ISEL) and Iressa NSCLC Trial Evaluating REsponse and Survival versus Taxotere (INTEREST). Although the phase III ISEL trial failed to prove the superiority of gefitinib treatment compared to placebo in previously treated patients, a subgroup analysis demonstrated improved survival in particular populations (Asians and non-smokers). The INTEREST study compared an EGFR tyrosine kinase inhibitor with chemotherapy in pretreated advanced non-small-cell lung cancer. In INTEREST, survival was similar for gefitinib and docetaxel in almost all subgroups; no EGFR-related biomarker or any clinical factor (including female sex, adenocarcinoma histology, never-smoker, and Asian ethnicity) appeared to be predictive of a greater survival benefit for gefitinib versus docetaxel. However, these factors may still be predictive of a greater survival benefit for gefitinib and/or docetaxel versus best supportive care; alternatively, they may just be good prognostic factors. Progression free survival and overall response rate was no statistically significant difference between gefitinib and docetaxel. This suggests gefitinib can provide similar overall survival to docetaxel in pretreated advanced non-small-cell lung cancer patients. These studies have demonstrated that gefitinib is effective for the second-line treatment of NSCLC. Now, gefitinib is recommended in advanced and metastatic NSCLC as second-line chemotherapy.

But, there was no prospective study with gefitinib in NSCLC wih squamous cell histology. This trial will investigate the efficacy and safety of gefitinib in locally advanced, metastatic NSCLC patients with squamous cell histology who have failed first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced(stage IIIB or IV) squamous NSCLC
2. Failure of only one first line chemotherapy for advanced disease
3. At least one lesion that unidimensionally measurable by computed tomography (RECIST 1.1)
4. Performance status: ECOG 0-2
5. Age ≥20
6. Adequate renal function: serum creatinine level < 2 mg/dL (177 μmol/L)
7. Adequate liver functions

   * : Transaminase (AST/ALT) < 2 X upper normal value
   * Bilirubin < 2 X upper normal value
8. Adequate hematological function: hemoglobin ≥ 9 g/dL absolute neutrophil count (ANC) ≥ 1,500/μL and platelet count ≥ 100,000/μL
9. Life expectancy 3 months
10. Written Informed consent prior to any study specific procedures
11. NSCLC with an activating sensitizing EGFR mutation

Exclusion Criteria:

1. Two or more chemotherapy treatment regimen for advanced disease
2. Previous therapy with other EGFR-TKI related drug
3. Known or suspected brain metastases or spinal cord compression
4. Radiotherapy within 4 weeks before study entry
5. Any other malignancies within the past 5 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
6. Pregnant or lactating women
7. Other serious illness or medical conditions as judged by the investigator
8. Known severe hypersensitivity to gefitinib or any of the excipients of the product
9. Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy.
10. Presence of EGFR mutation reported to confer resistance to EGFR TKI: exon 20 point mutation (T790M or S768I EGFR) or exon 20 insertion
11. Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy.
12. Concomitant use of known CYP 3A4 inducers such as phenytoin, carbamazepine, rifampicin, barbiturates,
13. Involvement in the planning and/or conduct of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-10; Primary Completion 2011-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Disease control rate (complete response, partial response, or stable disease) at 8 weeks | 8 weeks

SECONDARY OUTCOMES:
number of participants with adverse events as a measure of safety and tolerability | 2 years
  safety & tolerability: NCI CTCAE version 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Bong-Seog Kim, M.D, Principal Investigator — Seoul Veterans Hospital
Locations (1):
- Seoul Veterans Hospital, Seoul, South Korea